CLINICAL TRIAL: NCT05334095
Title: Angio-seal VIP Versus Perclose ProGlide for Closure of the Femoral Artery in Peripheral Vascular Disease: a Prospective Single-center Randomized Non-inferiority Trial
Brief Title: Angio-seal VIP Versus Perclose ProGlide for Closure of the Femoral Artery in Peripheral Vascular Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiongjing Jiang (Other)
Responsible Party: Sponsor-Investigator, Xiongjing Jiang, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-ZX09
Record Dates: First submitted 2022-04-06; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Peripheral Vascular Diseases; Percutaneous Intervention Via Femoral Artery
Keywords: Peripheral Vascular Diseases; closure device; Femoral Artery
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Perclose ProGlide (Active Comparator): Perclose ProGlide 6F Suture-Mediated Closure (SMC) System
  Interventions: Device: Perclose ProGlide
- Angio-seal VIP (Placebo Comparator): Angio-seal VIP Vascular Closure Device
  Interventions: Device: Angio-seal VIP

INTERVENTIONS:
Device: Perclose ProGlide — After peripheral vascular diagnostic and interventional procedures, patients are randomized to receive Perclose ProGlide.
  Arms: Perclose ProGlide
Device: Angio-seal VIP — After peripheral vascular diagnostic and interventional procedures, patients are randomized to receive Angio-seal VIP
  Arms: Angio-seal VIP

SUMMARY:
This study is designed to evaluate the efficacy (device deployment characteristics and performance) and safety (adverse access site related events) of Perclose ProGlide (Abbott Vascular Devices) for femoral access site closure in patients undergoing peripheral vascular diagnostic and interventional procedures in comparison with Angio-seal VIP (St. Jude Medical).

DETAILED DESCRIPTION:
Prospective, single-center, randomized (1:1), open-label, non-inferiority study in 1062 patients comparing Perclose ProGlide (test device) to the Angio-seal VIP (standard comparator).

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥18 and < 85 years of age.
* Patient is willing to provide written informed consent prior to study device use.
* Patient is undergoing a peripheral vascular diagnostic and/or interventional procedure via femoral arterial access.
* Patients' arterial puncture site is in the common femoral artery confirmed by a femoral angiogram, and ≥10mm away from the ostium of the inferior epigastric artery (IEA) and the bifurcation of superficial femoral artery and the profunda femoris artery.

Exclusion Criteria:

* The femoral access site has been punctured within 30 days, or deployed with a collagen-based hemostasis device within 90 days, or a suture-mediated closure device.
* Patients having a hematoma, pseudoaneurysm or arteriovenous fistula present prior to sheath removal confirmed by a femoral angiogram.
* Patients with minimum femoral artery calcium which is fluoroscopically visible at access site or femoral artery diameter stenosis greater than 50%.
* Ankle-brachial index (ABI) of the ipsilateral limb of access site cannot be measured due to severe peripheral artery disease (PAD).
* Patients who are pregnant or lactating.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1062 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of the device successfully deployed and absence of the major vascular complications necessitating aggressive treatments (surgical or percutaneous repair etc.) at 30 days | 30 days post procedure
  Deployment procedure success is defined as haemostasis after the delivery and release of a closure device, manual compression is no longer needed or less than 5 minutes, and no more closure devices are needed.
  Major vascular complications include:
  1. Vascular injury related to access site requiring surgical or percutaneous intervention, or ultrasound guided compression, or thrombin injection.
  2. New onset lower extremity ischemia attributed to arterial access or closure, and/or the ABI of the ipsilateral limb of access site decreased by ≥0.15 or requiring surgical or additional percutaneous intervention.
  3. haemorrhage related to access site requiring transfusion, or haemoglobin decreased by ≥5g/dl or hematocrit (HCT) decreased by ≥15%
  4. Infection requiring a hospitalization extended for more than 24 hours or a new hospitalization or treatment with intravenous antibiotics.
  5. Nerve injury related to access site which is permanent or requires surgery.

SECONDARY OUTCOMES:
Minor ipsilateral access site complications at 30 days and generally no aggressive treatment is required | 30 days post procedure
  Minor ipsilateral access site vascular complications included:
  1. Access site pseudoaneurysm or AV fistula documented by ultrasound, neither surgical nor percutaneous intervention is required.
  2. Post-discharge access site-related haemorrhage requiring ≥ 30 minutes manual compression to re-achieve hemostasis.
  3. Lower extremity arterial stenosis attributed to arterial access or closure, whereas neither surgical nor percutaneous intervention is required.
  4. haemorrhage related to access site with no transfusion required. while, transfusion is required when haemoglobin decreased by <5g/dl or hematocrit (HCT) decreased by <15%.
  5. Access site hematoma ≥ 6 cm, neither blood transfusion nor surgical intervention is required.
  6. Localized access site infection treated with intramuscular or oral antibiotics.
  7. Transient access site-related nerve injury.
Incidence at 180 days of the composite endpoint of major vascular complications necessitating aggressive treatments (surgical or percutaneous repair etc.) | 180 days post procedure
  Major vascular complications include:
  1. Vascular injuries related to access site requiring surgical or percutaneous intervention, or ultrasound guided compression, or thrombin injection.
  2. New onset lower extremity ischemia that is attributed to arterial access or closure, and the ABI of the ipsilateral limb of access site decreased by ≥0.15 or requiring surgical or additional percutaneous intervention.
  3. Bleeding related to access site requiring transfusion or haemoglobin decreased by ≥5g/dl or hematocrit (HCT) decreased by ≥15%
  4. Infection requiring a extended hospitalization for more than 24 hours or a new hospitalization or treatment with intravenous antibiotics.
  5. Nerve injury related to access site is permanent or requires surgery.
Deployment procedure time | within 24 hours of device deployment
  Deployment procedure time was defined as elapsed time from the first skin break to final closure (skin to skin time)
Time to haemostasis from removing the sheath until haemostasis | within 24 hours of device deployment
  Haemostasis is considered as insignificant bleeding on the bandage or small continuous oozing, manual compression is no longer needed or less than 5 minutes.
Patients' comfort level during the deployment of the closure device using the visual analog scale (VAS) | within 5 minutes of device deployment
  0 cm means no pain, while 10 cm means the worst imaginable pain or the worst pain one had experienced

CONTACTS AND LOCATIONS:
Overall Officials: Xiongjing Jiang, MD, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Disease
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China